CLINICAL TRIAL: NCT02724969
Title: A Mobile, Semi-automated Text Message-based Intervention to Prevent Perceived Low or Insufficient Milk Supply
Acronym: MILK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Jill R. Demirci, PhD, RN, IBCLC, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO16020007; 5R00NR015106 (NIH)
Record Dates: First submitted 2016-02-08; First posted 2016-03-31 (Estimated); Results first posted 2023-02-21 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Feeding
Keywords: text messaging; short message service
MeSH Terms: conditions — Breast Feeding | interventions — Milk

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Lactation consultant providing assistance has no knowledge of group assignment. Statistician completing final analysis of data will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MILK intervention group (Experimental): Semi-automated text messages sent to participants' cellular phones 3-5 times per week beginning Week 25 of pregnancy, through 8 weeks postpartum, specific to breastfeeding support and prevention of perceived insufficient milk supply.
  Interventions: Behavioral: MILK or Text4Baby text message intervention
- Text4Baby control intervention group (Active Comparator): Text4Baby automated texts sent to participants' cellular phones 3-5 times per week from Week 25 of pregnancy through the postpartum period from the national Text4Baby system. Messages provide general prenatal and postpartum support, including breastfeeding.
  Interventions: Behavioral: MILK or Text4Baby text message intervention

INTERVENTIONS:
Behavioral: MILK or Text4Baby text message intervention — MILK text message intervention encompasses prenatal and postpartum breastfeeding support and education text messages. Text4Baby text message intervention encompasses prenatal and postpartum text messages about pregnancy, infant care, and postpartum issues.

SUMMARY:
The purpose of this pilot randomized trial is to determine the effectiveness, feasibility, and acceptability of a mobile, semi-automated text message-based intervention (MILK) to prevent perceived low or insufficient milk supply (PIM) among mothers without prior breastfeeding experience. PIM is the leading cause of premature breastfeeding cessation, and prior work shows that it is often rooted in low breastfeeding self-efficacy and misconceptions about lactation physiology and trajectory. The MILK intervention is designed to address PIM, as well as other common breastfeeding problems via semi-automated text messages of prenatal and postpartum breastfeeding education and support. Messages are time-sensitive (e.g., specific to gestational age, time since delivery) and based on the Breastfeeding Self-Efficacy (Social Cognitive) Theory; they are also modeled from pilot work that investigated how first-time mothers view, manage and describe breastfeeding problems. Messages were vetted with clinical lactation experts, as well as pregnant and postpartum women with no other children.

The MILK intervention will be trialed against a control intervention group, who will receive general perinatal education through the national Text4Baby system. The investigators will recruit approximately 186 healthy, pregnant women at 13-25 weeks gestation from Magee Women's Hospital clinics and outpatient sites. Women will be randomized via computer-generated simple randomization to the experimental or control intervention. Both groups will receive text messages 3-5 times per week from week 25 of pregnancy through week 8 postpartum. Measured outcomes of interest will include perceived breast milk supply, breastfeeding confidence, maternal anxiety, breastfeeding exclusivity, and breastfeeding duration. Data will be collected at baseline (13-25 gestational weeks), 34-36 gestational weeks, and at 1, 2, 4, and 8 weeks postpartum via online survey or telephone call. To assess the potential longer-term impact of the intervention, breastfeeding continuation and exclusivity will be reassessed via telephone at 6 months postpartum. Between group and group x time differences in outcome measures will be examined graphically and via linear mixed modeling. To inform modifications to MILK, telephone interviews will be conducted with a subset of participants in each group to assess and compare intervention use, burdens and challenges, and suggested alterations (8 weeks).

DETAILED DESCRIPTION:
The purpose of the MILK Trial is to examine and compare the effectiveness, feasibility, and acceptability of a semi-automated, text-based, theory-driven intervention ("MILK" intervention) to prevent perceived insufficient milk and its potential inter-related sequelae, including maternal anxiety and early breastfeeding cessation, among mothers without breastfeeding experience who intend to exclusively or nearly exclusively breastfeed. Specifically, the investigators will:

1. Determine the effect of the MILK intervention on perceived insufficient milk supply (PIM) and related maternal psychological and behavioral sequelae.

   Compared to the control intervention group ("Text4Baby"), the investigators hypothesize that MILK participants will have a perception of greater breast milk volume/supply, higher self-reported breastfeeding confidence, lower anxiety scores, and longer duration of exclusive breastfeeding.
2. Assess the feasibility of a semi-automated text-based PIM intervention (MILK) for mothers.

The investigators will compare characteristics of women who are and who are not eligible for, chose to participate in, and complete this randomized pilot intervention study. The investigators will also conduct post-study individual interviews with mothers to determine how the interventions were used and perceived (e.g., burden, challenges).

ELIGIBILITY:
Inclusion Criteria:

Pregnant women who:

1. are ≥ 18 years;
2. are between 13-25 gestational weeks;
3. have no prior breastfeeding experience or other living biological children;
4. have a personal cell phone with internet access and an unlimited text message plan; and
5. intend to exclusively, or nearly exclusively breastfeed (<2 ounces of artificial milk per day) for at least 2 months postpartum; (6) plan to deliver their infant at MWH.

Exclusion Criteria:

1. Maternal, fetal, or neonatal conditions or complications with the potential to physiologically compromise breastfeeding or milk supply (e.g., history of breast reduction surgery, infant cardiac defects, postpartum infant ventilator dependence);
2. current gestation of ≥ 1 fetus;
3. contraindications to breastfeeding as specified by the American Academy of Pediatrics (e.g., HIV+ status).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Demirci, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demirci JR, Suffoletto B, Doman J, Glasser M, Chang JC, Sereika SM, Bogen DL. The Development and Evaluation of a Text Message Program to Prevent Perceived Insufficient Milk Among First-Time Mothers: Retrospective Analysis of a Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Apr 29;8(4):e17328. doi: 10.2196/17328. PMID 32347815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between February 2017 and May 2018 at prenatal visits at a single academic medical center. Recruitment also occurred through local print advertising, a University research registry, and social media. The first participant was enrolled on February 10, 2017, and the last participant was enrolled on May 14, 2018.
Pre-assignment Details: Of 413 participants assessed for eligibility, 250 met eligibility criteria, agreed to participate, and were randomized to a treatment group.
Period: Overall Study
Arm/Group | MILK Intervention Group | Text4Baby Control Intervention Group
Started | 126 | 124
Completed | 111 | 113
Not Completed | 15 | 11
Not completed — Lost to Follow-up | 12 | 6
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Infant demise | 0 | 2

BASELINE CHARACTERISTICS:
Population: Measures with numbers analyzed less than the overall baseline numbers include all participants with data collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | MILK Intervention Group | Text4Baby Control Intervention Group | Total
Number analyzed (Participants) | 126 | 124 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.5) | 28.7 (5.2) | 28.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 124 | 250
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity assessed at baseline with n=247 participants' data available
  Participants
    number analyzed (Participants) | 124 | 123 | 247
    Hispanic or Latino | 3 | 7 | 10
    Not Hispanic or Latino | 120 | 116 | 236
    Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race assessed at baseline with n=247 participants' data available
  Participants
    number analyzed (Participants) | 124 | 123 | 247
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 7 | 5 | 12
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 25 | 22 | 47
    White | 87 | 94 | 181
    More than one race | 3 | 2 | 5
    Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 126 | 124 | 250
Married [Count of Participants; unit: Participants] — Population: marital status assessed at baseline with n=247 participants' data available
  Participants
    number analyzed (Participants) | 124 | 123 | 247
    (all) | 81 | 77 | 158
Education level [Count of Participants; unit: Participants] — Population: education assessed at baseline with n=247 participants' data available
  Participants
    number analyzed (Participants) | 124 | 123 | 247
    Highschool or less | 15 | 13 | 28
    Associate's degree, vocational degree, or some college | 25 | 31 | 56
    Bachelor's degree | 36 | 33 | 69
    Postgraduate degree | 48 | 46 | 94
Employed at enrollment [Count of Participants; unit: Participants] — Population: employment assessed at baseline with n=237 participants' data available
  Participants
    number analyzed (Participants) | 124 | 123 | 247
    (all) | 104 | 108 | 212
Special Supplemental Program for Women, Infants, and Children (WIC) recipient [Count of Participants; unit: Participants] — Population: WIC status assessed at baseline with n=246 participants' data available
  Participants
    number analyzed (Participants) | 123 | 123 | 246
    (all) | 32 | 28 | 60
Infant Feeding Intentions Scale Score at enrollment [Mean (Standard Deviation); unit: units on a scale] — Only items 3-5 included from Infant Feeding Intentions (IFI) Scale, as items 1-2 part of study eligibility (score range 0-12, with higher score indicative of stronger intention to exclusively breastfeed up to 6 months postpartum) Population: Scale administered at baseline with n=246 participants' data available
  units on a scale
    number analyzed (Participants) | 124 | 122 | 246
    (all) | 10.2 (2.3) | 10.5 (2.2) | 10.3 (2.2)
Breastfeeding Self-Efficacy Scale (Short Form) Score Baseline [Mean (Standard Deviation); unit: units on a scale] — Score range 14-70, with higher scores indicative of higher breastfeeding self-efficacy Population: Scale administered at baseline with n=247 participants' data available
  units on a scale
    number analyzed (Participants) | 124 | 123 | 247
    (all) | 48.0 (8.6) | 48.1 (8.9) | 48.1 (8.7)
Iowa Infant Feeding Attitude Scale [Mean (Standard Deviation); unit: units on a scale] — Score range 17-85, with higher scores indicative of more positive breastfeeding attitude Population: Scale administered at baseline with n=247 participants' data available
  units on a scale
    number analyzed (Participants) | 124 | 123 | 247
    (all) | 62.0 (6.2) | 62.6 (6.6) | 62.3 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Perception of Milk Supply
Description: Assessed via the H & H Lactation Scale (21-item Likert scale) Used items 11-20 (the PIBSS (Perceived Infant Breastfeeding Satiety Subscale) and the MIBSS (Maternal-Infant Breastfeeding Satisfaction Subscale); each item score 1-7, with total possible summative score 10-70; higher scores indicative of better outcome (lowered perception of insufficient milk); items 12-15 reverse scored
Time Frame: 8 weeks postpartum
Population: Not completed by participants who indicated they stopped breastfeeding prior to 8 weeks postpartum; if more than 2 items were not answered on scale, sum scale of score was not computed; if 2 items or less were missing, the missing item(s) score was computed with the mean item score for the scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MILK Intervention Group | Text4Baby Control Intervention Group
Number analyzed (Participants) | 98 | 93
score on a scale | 54.9 (13.0) | 56.2 (14.6)
Statistical Analysis 1: Comparison: MILK Intervention Group vs Text4Baby Control Intervention Group; Test type: Superiority; p = .272, Mixed Models Analysis

2. Secondary Outcome: Breastfeeding Self-efficacy
Description: assessed via 14-item Breastfeeding Self-Efficacy Scale (Likert scale) Score range 14-70, with higher scores indicative of higher breastfeeding self-efficacy
Time Frame: 8 weeks postpartum
Population: Not completed by participants who indicated they stopped breastfeeding prior to 8 weeks postpartum; if no answer provided for more than 2 items in scale, scale score not computed and considered missing data. If < 2 items on scale incomplete, mean individual score on the other items was imputed for the missing value
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MILK Intervention Group | Text4Baby Control Intervention Group
Number analyzed (Participants) | 98 | 92
score on a scale | 51.8 (11.7) | 53.2 (12.2)
Statistical Analysis 1: Comparison: MILK Intervention Group vs Text4Baby Control Intervention Group; Test type: Superiority; p = .082, Mixed Models Analysis

3. Secondary Outcome: Maternal Anxiety and Depression
Description: 3-item PRAMS (Likert scale for each item 1-5; summative score range 3-15, with higher score indicative of greater depression and/or anxiety)
Time Frame: 8 weeks postpartum
Population: Not completed by participants who indicated they had stopped breastfeeding prior to 8 weeks postpartum
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MILK Intervention Group | Text4Baby Control Intervention Group
Number analyzed (Participants) | 104 | 99
score on a scale | 5.6 (2.3) | 5.2 (2.3)
Statistical Analysis 1: Comparison: MILK Intervention Group vs Text4Baby Control Intervention Group; Test type: Superiority; p = .355, Mixed Models Analysis

4. Secondary Outcome: Breastfeeding Continuation
Description: whether participant is doing any breastfeeding at 8 week assessment; dichotomous (yes/no); count represents "yes," participants indicating they are doing any breastfeeding at 8 weeks; abstracted from survey item assessing all feeding method(s) at 8 weeks
Time Frame: 8 weeks postpartum
Population: Only includes participants with breastfeeding data available at 8 weeks (i.e., participants who completed breastfeeding survey item(s) at 8 weeks or indicated they stopped breastfeeding prior to 8 weeks); note that some participants do not have 8 week breastfeeding data or 8 week survey data, but went on to complete the study by completing subsequent study timepoints
Measure: Count of Participants; unit: Participants
Arm/Group | MILK Intervention Group | Text4Baby Control Intervention Group
Number analyzed (Participants) | 112 | 112
Participants | 98 | 93
Statistical Analysis 1: Comparison: MILK Intervention Group vs Text4Baby Control Intervention Group; Test type: Superiority; p = .780, Mixed Models Analysis

5. Secondary Outcome: Breastfeeding Exclusivity
Description: whether participant is feeding 100% breast milk; dichotomous (yes/no), count represents "yes", exclusive breastfeeding/100% breast milk; abstracted from survey item assessing all feeding method(s) at 8 weeks
Time Frame: 8 weeks postpartum
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | MILK Intervention Group | Text4Baby Control Intervention Group
Number analyzed (Participants) | 112 | 112
Participants | 61 | 63
Statistical Analysis 1: Comparison: MILK Intervention Group vs Text4Baby Control Intervention Group; Test type: Superiority; p = .588, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: From study enrollment at 13-25 weeks of gestation until conclusion of the intervention and data collection of primary aims at 8 weeks postpartum
Description: Only reportable adverse events were collected/recorded for the study, and here we are only including reportable adverse events for maternal participants. Infants of participants are not included in numbers. Relevant to this, all-cause mortality does not include infants. As such, we report here that there were two infant deaths during the course of the study in the control group, and it was determined that they were unrelated to the study.
Arm/Group | MILK Intervention Group | Text4Baby Control Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/124
Other Adverse Events (participants affected / at risk) | 0/126 | 0/124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT02724969/Prot_SAP_ICF_000.pdf